CLINICAL TRIAL: NCT03977389
Title: Total Wrist Denervation: Survival Study and Functional Outcomes
Acronym: DTDPESERF
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: DTDPESERF (29BRC18.0122)
Record Dates: First submitted 2019-05-27; First posted 2019-06-06 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Wrist Arthritis; Survival
Keywords: Long-term result; Denervation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Population of the study: Patient undergoing total wrist denervation between January 1995 and December 2013 at Brest CHRU, performed by the same senior surgeon.
  Total wrist denervation is a routine procedure in orthopedic surgery for wrist arthritis.
  Interventions: Procedure: Total wrist denervation

INTERVENTIONS:
Procedure: Total wrist denervation — Study of the files

SUMMARY:
The purpose of the study is to evaluate the long-term effectiveness of total wrist denervation on pain by assessing the surgery survival.

The residual functional wrist's quality and the patients' satisfaction will also be evaluate.

DETAILED DESCRIPTION:
The degenerative diseases of the wrist are numerous and include both post-traumatic osteoarthritis lesions and inflammatory diseases. In any case, one of the main reasons for consultation is pain. In case of inefficiency of a well-conducted medical treatment (splints, anti-inflammatories, infiltrations), surgical management remains difficult because of the multitude of treatments that can be offered: partial or total arthrodesis of the wrist, prosthetic arthroplasties, pyrocarbon implants or proximal row carpectomy. But these treatments are heavy and can potentially be sources of complications such as stiffness, loss of strength or progressive wear of the implant.

Total wrist denervation is an alternative since 1966. The original technique follows an anatomical study of the innervation of the upper limb. This technique has been proven to significantly improve pain without major after effects. Several teams demonstrated a decrease in pain associated with conserved strength and mobility, but few studies have studied the long-term results of this technique, especially on the absence of residual pain.

The purpose of this study is to evaluate the long-term effectiveness of denervation on pain by assessing the surgery survival, the residual functional wrist's quality and the patients' satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* patient undergoing total wrist denervation between January 1995 and December 2013 at Brest CHRU, performed by the same senior surgeon

Exclusion Criteria:

* patient who had another intervention at the same time (confounding factor)
* refusal expressed by the patient to participate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing total wrist denervation (TWD) between January 1995 and December 2013 at Brest CHRU, performed by the same senior surgeon.
  TWD was indicated in a routine procedure for degenerative diseases of the wrist (post-traumatic osteoarthritis lesions and inflammatory diseases).
  The aetiologies are varied: SLAC-wrist, distal radius fractures, SNAC-wrist, Kienböck disease, chondrocalcinosis, peri-lunar luxation of the carpus, rheumatoid arthritis, haemochromatoses, ruptures of the luno-triquetral ligament.
Sampling Method: Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
survival over time | from date of surgery until the date of first documented failure (surgical revision; pain > 3), assessed up to the inclusion date
  duration (in years) of absence of surgical revision, and residual pain < or = 3 on a pain numerical scale (0 to 10, WHO criteria for mild pain)

SECONDARY OUTCOMES:
surgery survival over time | from date of surgery until the date of documented failure (surgical revision), assessed up to the inclusion date
  duration (in years) of absence of surgical revision
residual pain | at the inclusion date
  numeric pain rating scale (between 0 to 10; 0 equal no pain; 10 equal "worst pain imaginable")
residual functional wrist's quality | at the inclusion date
  Result of the DASH (Disabilities of the Arm and Shoulder Disabilities) score (between 0 to 100; 0 equal better result; 100 equal worst result)
patients' satisfaction (1) | at the inclusion date
  analogue scale between 0 to 10 at the last follow-up (0 equal minimum; 10 equal maximum)
patients' satsfaction (2) | at the inclusion date
  answer to "would you repeat this procedure again?"

CONTACTS AND LOCATIONS:
Locations (1):
- CHUR de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: No